CLINICAL TRIAL: NCT07276139
Title: Pacing Advancements With Cost and Experience VALuation for Unified Patient-Led Clinical Evidence - the PACEVALUE Study
Brief Title: PACEVALUE: Development of a Risk Score to Predict Pacing-Induced Cardiomyopathy in Patients Undergoing Pacemaker or ICD Implantation and Evaluation of Patient Outcomes and Cost-Effectiveness Across Different Healthcare Systems
Acronym: PACEVALUE
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-02109
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiomyopathy, Secondary; Arrhythmias, Cardiac; Heart Failure; Pacing Induced Cardiomyopathy; Conduction System Pacing
MeSH Terms: conditions — Cardiomyopathies; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PACEVALUE study is a large, international observational study aiming to improve the treatment of patients receiving cardiac implantable electronic devices (CIEDs) such as pacemakers, implantable cardioverter-defibrillators (ICDs), and cardiac resynchronization therapy (CRT) devices. While these devices are vital for managing heart rhythm disorders and heart failure, chronic right ventricular pacing can sometimes cause a condition called pacing-induced cardiomyopathy (PICM), where the left side of the heart weakens over time, leading to increased hospitalizations and higher mortality.

The main goal of the study is to develop and validate a risk prediction model using routine clinical and device data to identify patients at highest risk of PICM before device implantation. By stratifying patients according to this risk score, the study aims to guide personalized pacing strategies, including conduction system pacing (CSP) and CRT options, to improve outcomes and reduce complications.

The study will recruit approximately 4,500 patients across multiple centers in Europe and Australia, with planned future inclusion of sites in the UK. Participants will be followed for a minimum of two years, with data collection including heart function imaging, device data, clinical outcomes, patient-reported outcomes (PROMs/PREMs), and healthcare costs.

This observational study will also compare clinical practices and cost-effectiveness of different pacing strategies across diverse healthcare systems, aiming to inform evidence-based, patient-centered, and economically efficient device therapy decisions. The findings will lay the groundwork for future registry-based randomized controlled trials to further optimize pacing treatments.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to enrollment
* Age ≥18 years
* Undergoing a CIED implantation (permanent pacemaker, ICD, or CRT)
* Willing and able to participate in long-term follow-up
* Sufficient language comprehension (or support) to provide informed consent and complete PROMs/PREMs.

Exclusion Criteria:

* Severe cognitive impairment without a legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients undergoing CIED implantation for standard clinical indications. Participants are recruited from multiple international centers in Switzerland, Bulgaria, Croatia, Poland, Australia, and the UK. The population includes patients receiving pacemakers, ICDs, or CRT devices. Patients with existing CRT at baseline serve as a comparator. The study collects real-world clinical practice data, imaging, device parameters, and PROMs/PREMs during long-term follow-up. Enrollment reflects diverse healthcare settings and demographics.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants developing PICM, defined as an absolute decline in left ventricular ejection fraction (LVEF) of ≥10 percentage points to ≤50% during long-term follow-up after CIED implantation | up to 2 years after device implantation

SECONDARY OUTCOMES:
Number of participants who died from any cause on follow-up | up to 5 years after device implantation
Number of participants hospitalized for heart failure on follow-up | up to 5 years after device implantation
Number of participants hospitalized for other cardiovascular events (excluding heart failure) on follow-up | up to 5 years after device implantation
Number of participants hospitalized for non-cardiovascular reasons on follow-up | up to 5 years after device implantation
Number of participants undergoing upgrade to CRT on follow-up | up to 5 years after device implantation
Number of participants with device-related complications on follow-up | up to 5 years after device implantation
Change in EQ-5D-5L Index Score from Baseline (range 0-1; higher scores indicate better quality of life) | at Baseline, 8 weeks, 1, 2, 3, 4, and 5 years
Change in patient satisfaction score with remote monitoring from Baseline (range 0-10; higher scores indicate higher satisfaction) | Baseline, 8 weeks, 1, 2, 3, 4, and 5 years
Total healthcare costs per patient for CSP versus right ventricular pacing, applying the PICM risk prediction score | up to 5 years after device implantation
Incremental cost-effectiveness ratio (ICER) of CSP versus right ventricular pacing per quality-adjusted life year (QALY) gained, applying the PICM risk prediction score | up to 5 years after device implantation
Inter-center and inter-country variation in CIED practice, including percentage of patients receiving CSP | up to 5 years after device implantation
Average percentage of ventricular pacing on follow-up | up to 5 years after device implantation
Number of participants with device-detected subclinical atrial fibrillation on follow-up | up to 5 years after device implantation
Number of participants experiencing stroke, stratified by modified Rankin Score on follow-up | up to 5 years after device implantation
Number of participants with moderate or severe tricuspid valve regurgitation on echocardiography on follow-up | up to 5 years after device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Nikola A. Kozhuharov, PD Dr. med., Principal Investigator — Inselspital, University Hospital Bern, Clinic of Cardiology
Locations (1):
- Inselspital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided